CLINICAL TRIAL: NCT04129736
Title: Determination of Teriflunomide Concentration in Serum and Cerebrospinal Fluid From Patients With Multiple Sclerosis Treated With Teriflunomide 14 mg Daily.
Brief Title: Teriflunomide Concentration in Serum and Cerebrospinal Fluid From Patients With Multiple Sclerosis
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Jan Lycke (Other)
Responsible Party: Sponsor-Investigator, Jan Lycke, Professor, Sahlgrenska University Hospital
Organization: Sahlgrenska University Hospital (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TERIFL0519; 2016-004414-10 (EudraCT Number)
Record Dates: First submitted 2019-10-15; First posted 2019-10-17 (Actual); Last update posted 2022-12-12 (Actual); Status verified 2022-12

CONDITIONS: Multiple Sclerosis, Pharmacokinetics
MeSH Terms: conditions — Multiple Sclerosis | interventions — teriflunomide

STUDY DESIGN:
Intervention Model Description: Pharmacokinetic
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Teriflunomide 14 mg tablets (Other): Single arm
  Interventions: Drug: Teriflunomide 14 MG

INTERVENTIONS:
Drug: Teriflunomide 14 MG — Blood and cerebrospinal fluid is obtained from teriflunomide treated patients with multiple sclerosis

SUMMARY:
Serum and cerebrospinal fluid will be obtained from 20 patients with relapsing-remitting multiple sclerosis treated with teriflunomide tablets 14 mg daily

DETAILED DESCRIPTION:
Teriflunomide concentration in cerebrospinal fluid and serum will be determined in 12 patients with multiple sclerosis. They have been treated for at least 6 months and the sampling from blood and by spinal tap is done before dose at 8 am in 10 patients and at 12 am in 10 patients. The dependence from age, sex, and blood-brain barrier (BBB) integrity will be evaluated.The ratio between serum and cerebrospinal fluid will determine the passage over the BBB.

ELIGIBILITY:
Inclusion Criteria:

* patients with multiple sclerosis treated with teriflunomide 14 mg for at least 6 months

Exclusion Criteria:

* other immunosuppressive or immunomodulating drugs, other CNS diseases

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2019-10-10 (Actual); Primary Completion 2021-03-31 (Actual); Study Completion 2021-06-30 (Actual)

PRIMARY OUTCOMES:
Concentration of teriflunomide in cerebrospinal fluid | one year

CONTACTS AND LOCATIONS:
Locations (1):
- MS Centre, Gothenburg, Västra Götaland County, Sweden

IPD SHARING:
Plan to Share IPD: No
No additional plan will be added